



Mr Daniel Howgate

Honorary Specialty Registrar Trauma & Orthopaedic Surgery and DPhil Student Botnar Institute of Musculoskeletal Sciences, University of Oxford, Old Road, Oxford, OX3 7LD

E-mail: daniel.howgate@ndorms.ox.ac.uk Oxford telephone number: 01865 760063

| Study Code: | Site ID Code: | Patient identification number: | |
|---|---|---|---|
| _ | | | - |

## **PATIENT CONSENT FORM**

## **THR PERFORMANCE & ASSESSMENT**

| Nar | ne of Researcher: | | If you agree, please initial | box |
|---|---|---|---|---|
| 1. | I. I confirm that I have read the information sheet dated (version) for this study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | | | |
| 2. | . I understand the lead researcher and research team (supervisors or collaborators) will have access to the minimum personally-identifiable information possible. Only completely anonymised data will be used outside of NHS premises. | | | |
| 3. | 3. I understand that responsible members of the University of Oxford may be given access to anonymised study records data for monitoring and/or audit of the study to ensure that the research is complying with applicable regulations. | | | |
| 4. | 4. I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | | |
| 5. | . I agree to take part in this study. | | | |
| | ame of Participant | <br>Date | <br>Signature | |
| _ | | | | |
| Name of Person taking<br>Consent | | Date | Signature | Signature |
| THR | ent Consent form Performance & Assessment | | Version 2.0 12 <sup>th</sup> October 201<br>REC Reference number: 19/<br>IRAS Ref: 270167 | |

| *1 copy for participant; 1 copy for researcher site file; 1 | (original) to be kept in medical notes (if part | ticipant is a patient). |
|---|---|---|